CLINICAL TRIAL: NCT05360433
Title: Impact of Reduced Initial Prescription Size on Opioid Consumption in Postoperative Pain Management for Scheduled Cesarean Deliveries
Brief Title: Too Much of a Good Thing? Impact of Initial Prescription Size in Post-cesarean Section Pain Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jaclyn D Nunziato, Assistant Professor of Obstetrics and Gynecology, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-516
Record Dates: First submitted 2022-03-03; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
Keywords: cesarean section; opioid prescription; narcotics; opioids; post operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 10 tablet prescription group (Active Comparator): These participants receive 10 tablets of oxycodone 5 mg at discharge for postoperative pain.
  Interventions: Drug: Oxycodone oral capsule
- 20 tablet prescription group (Active Comparator): These participants receive 20 tablets of oxycodone 5 mg at discharge for postoperative pain.
  Interventions: Drug: Oxycodone oral capsule

INTERVENTIONS:
Drug: Oxycodone oral capsule — Reduced initial prescription of oxycodone for postoperative pain management following cesarean section.
  Other Names: opioid prescription size

SUMMARY:
This is a randomized controlled trial involving 170 opioid naive women ages 19-40 undergoing scheduled C-sections at Carilion Roanoke Memorial Hospital. Participants are randomized to receive either 10 or 20 tabs of oxycodone 5mg as an initial postoperative prescription in a double-blinded parallel trial design. Outcome metrics related to overall opioid consumption and patient satisfaction with pain management are collected at three different time points post-operative: 2-3 days (in hospital), 10-14 days, and 6 weeks.

DETAILED DESCRIPTION:
All faculty scheduled cesarean deliveries will be eligible for possible enrollment. Once patients are scheduled for delivery, their providers will grant permission for potential participation in the study. Two weeks prior to surgery, potential participants will receive a phone call to assess interest and eligibility for participation. During the phone call, investigators will explain the goals of this research project and the overall study design. If an individual expresses interest in participation during this initial phone call, investigators will administer an intake survey. The intake survey is designed to collect data on participant eligibility as well as preexisting attitudes and experiences that may influence postoperative opioid consumption.

Patients who complete the initial survey will be approached by a member of the research team on postoperative day two or three prior to discharge from the hospital. At this time, investigators will obtain informed consent and provide each participant with an enrollment packet prepared by the principal investigator. The enrollment packet will contain educational components including information about opioids with specific instructions about how to use opioids for pain management and instructions on proper disposal of unused tablets. Investigators will also include information about alternative forms of analgesia (ibuprofen and acetaminophen) with FDA approved instructions regarding their use in pain management. The study team's goal in including these educational components for each study group is to ensure that women are able to make safe and informed decisions regarding both forms of medication for optimal pain management. The enrollment packet will also include copies of all surveys the participants will be completing and a visual representation of the numerical pain scale for participants to reference.

Women in the study will be randomized to receive either 10 or 20 tablets of oxycodone 5 mg upon discharge. Randomization of prescription groups will be achieved using a computer randomized sequence assigning participants in a 1:1 ratio to either a standard discharge prescription size (20 tablets oxycodone 5mg) or a reduced initial prescription size (10 tablets oxycodone 5 mg). Participants will not be given information regarding prescription size of other participants in the study, and will therefore be blinded as to whether or not their prescription size represents the larger or smaller group.In the event that a participant should require more opioid tablets for pain medication, there will be an option to request a refill from a designated provider. Refills across both groups will be standardized to a size of 5 tablets and healthcare providers will be notified of the participant's request in order to help determine if an earlier postoperative visit is needed for evaluation.

Outcome metrics will be collected at 3 different postoperative time points. The initial "inpatient survey" will be completed in person at the time of consent on postoperative day two or three. This survey is designed to collect information about each participant's perceived pain experience during inpatient stay and capture pain rating at time of discharge. Outcome metrics at two subsequent time points (10-14 days post-op and 6 weeks post-op) will be collected using an "outpatient survey." Participants will be given the option to complete the outpatient surveys over the phone with the investigator directly inputting metrics or through an online survey directly linked to the study electronic database. Follow-up surveys will assess a number of outcome metrics related to opioid use, participant's pain experience, and participant satisfaction with pain management.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 19-40 years old
* Pregnant
* Scheduled to undergo cesarean section at Carilion Roanoke Memorial Hospital
* opioid naïve (defined as no opioid use within 30 days of surgery

Exclusion Criteria:

* History of chronic pain
* History of opioid use disorder
* History of any known intolerance or allergies to analgesics
* Women with postoperative complications (hysterectomy during or after birth, bowel or bladder injury during birth, need for re-operation, or immediate wound complication)
* Language barrier preventing screening or consent

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption by participants post-cesarean delivery | 2 weeks
  Number of tablets of oxycodone consumed for postoperative pain management. This will be measured by a pill count at the participant's 2 week post-op visit and the participant's responses to postoperative surveys at 2 weeks and 6 weeks post surgery.
Total opioid consumption by participants post-cesarean delivery | 6 weeks
  Number of tablets of oxycodone consumed for postoperative pain management. This will be measured by a pill count at the participant's 2 week post-op visit and the participant's responses to postoperative surveys at 2 weeks and 6 weeks post surgery.

SECONDARY OUTCOMES:
Participant pain rating | 2 weeks
  reported level pain based on Numeric Pain Rating Scale (NPRS) 0-10, with 0 being no pain and 10 being the worst pain imaginable
Participant pain rating | 6 weeks
  reported level pain based on Numeric Pain Rating Scale (NPRS) 0-10, with 0 being no pain and 10 being the worst pain imaginable
Participant satisfaction with pain management | 2 weeks
  Patient reported satisfaction with postoperative pain management on survey based on opinion of whether medications provided were strong enough and the quantity of medication provided Participants are asked "were you overall satisfied with your pain management since surgery" and answer yes or no
Participant satisfaction with pain management | 6 weeks
  Patient reported satisfaction with postoperative pain management on survey based on opinion of whether medications provided were strong enough and the quantity of medication provided Participants are asked "were you overall satisfied with your pain management since surgery" and answer yes or no
Requests for opioid prescription refills by participants | 2 weeks
  Number of opioid refills required by participant requesting additional medication up to 6 weeks post operative
Requests for opioid prescription refills by participants | 6 weeks
  Number of opioid refills required by participant requesting additional medication up to 6 weeks post operative

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn D Nunziato, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.